CLINICAL TRIAL: NCT00276081
Title: A Randomized Trial of Gabapentin, Estrogen and Placebo for the Treatment of Postmenopausal Hot Flashes
Brief Title: Gabapentin Versus Estrogen for the Treatment of Hot Flashes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO3 HD042609 NIH/NICHD; R03HD042609 (NIH)
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-01

CONDITIONS: Hot Flashes
Keywords: Hot flashes; postmenopausal; climacteric symptoms; hormone replacement therapy; gabapentin
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin; Estrogens

INTERVENTIONS:
Drug: Gabapentin, Estrogen and placebo administration

SUMMARY:
To compare the efficacy and safety of gabapentin, estrogen and placebo in the treatment of hot flashes and other climacteric symptoms.

DETAILED DESCRIPTION:
HRT is associated with an increased risk of thrombo-embolic events, breast cancer and cardiovascular events. Safe, effective, and well-tolerated alternative therapies for hot flashes are needed. Gabapentin is a gamma-aminobutyric acid (GABA)-analog that we have reported is associated with a reduction in the frequency of hot flashes in postmenopausal women who were taking gabapentin for other indications. However, it is not known whether the efficacy of gabapentin in the treatment of hot flashes and other menopausal symptoms is comparable to that of estrogen, the gold standard. For this study, 60 subjects are to be recruited and randomized into 3 arms of 20 each (gabapentin, estrogen and placebo).We will perform an analysis of the results after all 60 subjects have been recruited, screened, enrolled and completed the study. The investigators of the study continue to be blinded to the study groups and their randomization. To determine if gabapentin approaches the efficacy of estrogen in the treatment of hot flashes,postmenopausal women between ages 35 and 60 with 7-20 moderate-severe postmenopausal hot flashes/day will be randomized into a double-blinded placebo controlled trial of estrogen, gabapentin and placebo. All patients must meet stringent inclusion and exclusion criteria. Pre- and post-study hot flash diaries, depression and climacteria scales will be collected. Patients are required to undergo physical examination and blood work and to complete a daily hot flash and medication compliance records. Hot flash frequency and composite score for hot flashes will be calculated for the three groups based on the hot flash diary. Side effects, climacteric scale and depression scales will also be used.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal women between ages 35-60
2. Must experience 7-20, moderate-severe hot flashes/day or 50-140 moderate-severe hot flashes/week for greater than two months
3. Must have had a bilateral salpingo-oopherectomy for >12 months or amenorrhea>6 months or #4 (below)
4. Has an FSH>30 mIU/ml
5. Must have a signed informed consent
6. Able to function independent in all activities of daily living and be capable of reliable documentation

Exclusion Criteria:

1. Any contraindication to estrogen and progesterone replacement therapy
2. History of an MI, stroke, and/or functional decline.
3. Fails to record data in the hot flash diary>3 days during the 2 week baseline period.
4. Unable or willing to make required visits at the specified times over the course of therapy.
5. History of any malignancies or undiagnosed vaginal bleeding.
6. History of chronic liver, gallbladder, chronic renal, cardiac or endocrine diseases

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2002-05; Study Completion 2004-09

PRIMARY OUTCOMES:
Reduction in hot flash frequency

SECONDARY OUTCOMES:
Side effects
Effect on climacteric symptoms
Effect on depression

CONTACTS AND LOCATIONS:
Overall Officials: Sireesha Y. Reddy, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] Reddy SY, Warner H, Guttuso T Jr, Messing S, DiGrazio W, Thornburg L, Guzick DS. Gabapentin, estrogen, and placebo for treating hot flushes: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):41-8. doi: 10.1097/01.AOG.0000222383.43913.ed. PMID 16816054